CLINICAL TRIAL: NCT00004778
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Antenatal Thyrotropin-Releasing Hormone in Pregnant Women With Threatened Premature Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Children's Hospital of Philadelphia (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11826; CHP-92536
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Respiratory Distress Syndrome
Keywords: cardiovascular and respiratory diseases; neonatal disorders; rare disease; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Tract Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — Betamethasone; Dexamethasone; Thyrotropin-Releasing Hormone

INTERVENTIONS:
Drug: betamethasone
Drug: dexamethasone
Drug: thyrotropin-releasing hormone

SUMMARY:
OBJECTIVES: I. Evaluate the effect of thyrotropin-releasing hormone (TRH) on the severity of initial lung disease and occurrence of chronic lung disease when given antenatally to women with threatened premature delivery.

II. Evaluate possible mechanisms for the effects of TRH on the severity and incidence of chronic lung disease.

III. Investigate whether a deficiency in endogenous cortisol and/or thyroid hormones after birth influences the severity of lung disease and the development of chronic lung disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Participants are stratified by participating institution.

Participants are randomly assigned to 1 of 2 treatment groups. The first group is treated with intravenous thyrotropin-releasing hormone (TRH) and intramuscular injections of betamethasone or dexamethasone. The second group receives a placebo in place of TRH.

Postnatal therapy with surfactants, prophylactic steroids, and indomethacin is allowed.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Threatened premature delivery at 24 to 30 weeks gestation, i.e.: Premature labor Premature rupture of membranes Elective premature delivery medically indicated Fetal lung maturity immature or unknown --Prior/Concurrent Therapy-- No more than 72 hours since any initial corticosteroids --Patient Characteristics-- The following complications exclude: Fetal distress Amnionitis Severe maternal bleeding uncontrolled with transfusion or volume replacement Fetal or maternal heart disease Significant fetal blood loss Maternal blood pressure 140/90 mm Hg or higher with or without treatment Maternal hyperthyroidism Maternal hyperprolactinemic condition Significant fetal anomaly Multiple gestation with demise of 1 or more fetuses Nonimmune hydrops No participation in other clinical research projects

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1090
Dates: Start 1993-08

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A. Ballard, Study Chair — Children's Hospital of Philadelphia